CLINICAL TRIAL: NCT02713022
Title: Body Composition and White Adipose Tissue Inflammation
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-235
Record Dates: First submitted 2016-03-11; First posted 2016-03-18 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Prostate Cancer; Body Composition; White Adipose Tissue Inflammation
Keywords: DEXA Scan; 15-235
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Breast Cancer: DEXA scan will be carried out 1 to 30 days prior to mastectomy. Patients will also complete the Godin Leisure Time Exercise Questionnaire (GLTEQ) and their waist to hip ratio will be measured.
  Interventions: Device: DEXA Scan; Behavioral: Godin Leisure Time Exercise Questionnaire (GLTEQ)
- Prostate Cancer: DEXA scan will be carried out 1 to 30 days prior to radical prostatectomy. Patients will also complete the Godin Leisure Time Exercise Questionnaire (GLTEQ) and their waist to hip ratio will be measured.
  Interventions: Device: DEXA Scan; Behavioral: Godin Leisure Time Exercise Questionnaire (GLTEQ)

INTERVENTIONS:
Device: DEXA Scan
Behavioral: Godin Leisure Time Exercise Questionnaire (GLTEQ)

SUMMARY:
The investigators want to find a better way to predict the risk of having fatty tissue inflammation by using a different approach to finding out body fat composition. In this study, the investigators want to estimate the body fat composition using a DEXA scan. DEXA stands for dual energy X-ray absorptiometry. It is the standard and established test to determine bone mineral density (how strong the bones are) to diagnose osteoporosis. This test can also be used to determine the body composition including percent body fat and lean mass. The investigators will compare the participants DEXA scan results for body fat composition to the inflammation found in the breast tissue from the mastectomy to see if there is a relationship. If successful, this may help us predict which patients may be at risk for breast cancer in the future. In addition, the investigators will compare the participants DEXA scan results for body fat composition and inflammation found in the fat tissue from the mastectomy or prostatectomy to the level of exercise activity as measured by a short questionnaire to see if there is a relationship. The investigators will also measure the participants waist to hip ratio.

Finally, at the time the participant has blood drawn for their standard presurgical testing, the investigators will also test the blood for prediabetes using a blood test called hemoglocin A1c. The investigators will also measure for the participants waist to hip ratio, and a Hgb A1c blood drawn will be take at the time of presurgical testing. If not feasible, Hgb A1c can be drawn at a separate visit prior to the DEXA scan. If successful, this may help us predict which patients may be at risk for breast cancer in the future.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Female
* All BMIs
* Patients undergoing mastectomy at MSKCC (i.e. Nipple-sparing mastectomy, skin-sparing mastectomy, simple mastectomy, modified radical mastectomy, radical mastectomy); mastectomy may be either prophylactic or therapeutic. OR
* Patients undergoing hysterectomy at MSKCC
* History of prior breast surgeries/procedures is acceptable

Exclusion Criteria:

* Pregnancy (confirmed or suspected);
* Inability to lay supine on equipment table and maintain the position for the necessary time;
* Weight superior to the maximum allowed by the DEXA machine (over 350 lbs or 158 kg);
* Greater than 10% baseline weight loss in the past year;
* Planned surgical procedure is not a Mastectomy (i.e. breast conservation surgery or other non-mastectomy procedure; such as lumpectomy) or hysterectomy
* Metastatic cancer
* History of Wasting Syndromes or Cachexia
* Use of daily NSAIDs, aspirin, or steroids (other than inhaled or topical) within 30 days of surgery
* Use of neoadjuvant systemic or radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is open to patients undergoing prophylactic or therapeutic mastectomy or radical prostatectomy at MSKCC.
  Patients will be identified and recruited from the Breast Service at and Plastics and Reconstructive Surgery Clinics MSKCC and approached at the time of initial surgical consultation.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
fat percentage | 1 year
  as measured by DEXA
presence of White Adipose Tissue Inflammation (WATi ) | 1 year
  as measured by DEXA

CONTACTS AND LOCATIONS:
Overall Officials: Neil Iyengar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Waters Corporation (Data Analysis Only), Milford, Massachusetts
  - Memorial Sloan Kettering Cancer Center (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Weill Medical College of Cornell University (Data and Specimen Analysis Only), New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org